CLINICAL TRIAL: NCT04454450
Title: Integration of Radiomic Analysis Into the Multi-Modal Profiling of High-Grade Serous Ovarian Cancer
Brief Title: Using Advanced Imaging Studies to Develop a Profile of High-grade Serous Ovarian Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-212
Record Dates: First submitted 2020-06-23; First posted 2020-07-01 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Ovarian Cancer; High Grade Ovarian Serous
Keywords: FIGO stage IIIC-IV; PET radiotracer; 20-212
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Imaged prior to primary debulking surgery (Experimental): Imaging will include research PET/MRI of pelvis within 30 days of multiregion tissue collection. Concretely, in patients triaged to primary debulking surgery (PDS), PET/MRI will be obtained within 30 days preceding multi-region tissue collection at the time of PDS (already being done under IRB# 06-107).
  Interventions: Diagnostic Test: PET/MRI; Diagnostic Test: Contrast enhanced CT
- Imaged pre/postneoadjuvant chemotherapy (NACT) (Experimental): In patients triaged to neoadjuvant chemotherapy (NACT) and interval debulking surgery (IDS), PET/MRI will be obtained at two time points, i.e. first within 30 days preceding NACT/ multi-region laparoscopic tissue sampling (already being done under IRB# 06-107) and, second, any time after completion of NACT and before multi-region tissue collection at the time of interval debulking surgery (already being done under IRB# 06-107).
  Interventions: Diagnostic Test: PET/MRI; Diagnostic Test: Contrast enhanced CT

INTERVENTIONS:
Diagnostic Test: PET/MRI — Imaging will include research PET/MRI of pelvis within 30 days of multiregion tissue collection.For research PET/MRI - standard volumes of gadolinium contrast and fluorodeoxyglucose (FDG) will be administered.
Diagnostic Test: Contrast enhanced CT — Standard of care contrast enhanced CT

SUMMARY:
The researchers are doing this study to find out whether the researchers can combine information provided by PET/MRI scans with information from tests on blood and tissue samples to develop a very detailed description (profile) of high-grade serous ovarian carcinoma (HGSOC), which could improve our ability to treat this disease.

The study researchers will use computers to analyze the combined results of the imaging tests and the genetic and immune system tests on the tumor samples. The study researchers think that this information will help them more accurately predict the way tumors respond to treatment, which may improve their ability to individualize treatments for this disease.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age or older
* Histologically confirmed or clinically suspected FIGO stage IIIC-IV HGSOC
* Signed consent to MSK Institutional tissue banking protocol IRB# 06-107 and signed or planned to sign IRB# 12-245, and planned to undergo multi-region tissue collection [under the above IRB protocols] and plan to undergo subsequent tissue analysis under biospecimen IRB# 15-200.
* Staging standard-of-care contrast-enhanced CT of abdomen and pelvis (+/-chest) available in picture archiving and communication system (PACS) that was obtained at our institution as a part of standard-of-care work-up or submitted for from the outside
* Plasma glucose ≤200 mg/dL
* Negative pregnancy test, if a patient is of child-bearing potential

Exclusion Criteria:

* Known allergy to gadolinium-based contrast medium requiring premedication or known adverse reactions to gadolinium-based contrast medium.
* Known history of impaired renal function, with documented eGFR <30 within 30 days prior to PET/MRI.
* Patients who cannot give valid informed consent because of general medical or physical condition, or physiologic status unrelated to presence of ovarian cancer
* Patients who are unwilling or unable to undergo PET/MRI including patients with absolute or relative contraindications to MRI including breast tissue expanders, cardiac pacemakers and defibrillators, non MRI-compatible aneurysm clips, neurostimulators, programmable CSF shunts, vascular stents, claustrophobia, or inability to lie flat for the duration of the examination.
* Patients with metallic hardware, implant, or device in the abdomen or pelvis that might distort the local magnetic field and compromise image quality.
* Radiotherapy to the abdomen or pelvis within 12 months of the screening visit.
* Subjects with a current diagnosis of ovarian cancer other than HGSOC
* Patients with known synchronous primary endometrial cancer or past history of endometrial cancer.
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor. Patients may have received prior adjuvant chemotherapy for breast cancer.
* With the exception of non-melanoma skin cancer and other specific malignancies as noted above, subjects with excluded known concurrent malignancy.
* Unresolved bowel obstruction.
* History or current evidence of any condition, therapy, or lab abnormality that might confound the results of the study or interfere with patient's participation for the full duration of the study.
* Absence of any target lesions ( ≥1-2 cm) in the pelvis (right adnexa, left adnexa, infra-colic omentum, pelvic peritoneum) visible on staging standard-of-care CE-CT and accessible for tissue sampling at laparoscopy and/or primary/ interval debulking surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Ovarian Cancer
Enrollment: 10 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Comparison between radiologist tumor segmentation | 1 year
  Radiologist-defined tumor volumes will be used to train and validate a machine learning algorithm for generating segmentations. The data will be split into 70%-30% of training and test sets, respectively. The comparisons will be performed on a slice-by-slice and lesion-bylesion basis, which should ensure sufficient numbers of examples for testing.

CONTACTS AND LOCATIONS:
Overall Officials: Viktoriya Paroder, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm